CLINICAL TRIAL: NCT04008849
Title: A Follow-Up Study to Evaluate the Safety and Clinical Outcomes of Patients With Non-Malignant Disease Who Have Undergone Hematopoietic Stem Cell Transplantation With MGTA-456
Brief Title: A Follow-up Study in Patients With Inherited Metabolic Disorders (IMD) Who Underwent Hematopoietic Stem Cell Transplantation (HSCT) With MGTA-456
Acronym: IMD-002
Status: Terminated | Type: Observational
Why Stopped: Due to low enrollment
Sponsor: Magenta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IMD-002
Record Dates: First submitted 2019-05-23; First posted 2019-07-05 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Inherited Metabolic Disorders (IMD)
Keywords: Inherited Metabolic Disorders; Hematopoietic Stem Cell Transplant; MGTA-456; Umbilical Cord Blood Transplant; Hurler Syndrome; Cerebral Adrenoleukodystrophy; Globoid Cell Leukodystrophy; Metachromatic Leukodystrophy
MeSH Terms: conditions — Mucopolysaccharidosis I; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic | interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells & plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects treated with MGTA-456: MGTA-456 is an investigational expanded CD34+ cell therapy
  Interventions: Other: Safety and efficacy assessments

INTERVENTIONS:
Other: Safety and efficacy assessments — Long term safety and clinical outcomes

SUMMARY:
A follow-up study to evaluate the safety and clinical outcomes of patients with inherited metabolic disorders (IMD) who have undergone hematopoietic stem cell transplantation (HSCT) with MGTA-456

DETAILED DESCRIPTION:
This is a follow-up study to evaluate the long-term safety and efficacy outcomes of patients with inherited metabolic disorders (IMDs) who received MGTA-456 for HSCT in the core study. MGTA-456 is an expanded CD34+ cell therapy product candidate given after myeloablative conditioning to induce rapid and sustained hematopoietic engraftment. In patients with selected IMDs, transplant is expected to replace defective or missing protein, and preserve neurodevelopment. Patients with Hurler syndrome (also referred to as mucopolysaccharidosis-1H (MPS-1H)), cerebral adrenoleukodystrophy (cALD), metachromatic leukodystrophy (MLD) or globoid cell leukodystrophy (GLD) enrolled in the core study will be eligible to participate in this follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee-approved written informed consent form must be signed and dated by the patient or legal guardian. Study assents will also be prepared for children and adolescents to review when applicable.
* Patient completed an IMD study in the MGTA-456 program and was administered MGTA-456 for HSCT.

Exclusion Criteria:

•Patients enrolled in an IMD study in the MGTA-456 program who did not receive MGTA-456 or were withdrawn from the core study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects with an inherited metabolic disorder (IMD) that were treated with MGTA-456
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of related adverse events | 2 years
Incidence of serious adverse events | 2 years
Incidence of late hematological graft failure | 2 years
Incidence of chronic graft versus host disease | 2 years
Overall survival | 2 years
Event-free survival | 2 years
Change in cALD Neurologic Function Score over time | 2 years
Proportion of subjects without gadolinium enhancement on MRI over time | 2 years
Alpha-iduronidase blood enzyme level (nmol/hr/mg) in Hurler patients | 2 years
Very long chain fatty acid blood level (ug/mL) in cALD patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Orchard, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No